CLINICAL TRIAL: NCT02094027
Title: The Role of Self-help in the Pre-surgical Treatment of Binge Eating Disorder in Bariatric Surgery Candidates: Implications for Weight-related and Psychological Outcome.
Brief Title: Bariatric Surgery and Guided Self-help for Binge Eating Disorder
Acronym: BED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New evidence came to light to indicate that study was no longer relevant
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10/H0707/67
Record Dates: First submitted 2014-03-05; First posted 2014-03-21 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2014-03

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Binge eating; Self help
MeSH Terms: conditions — Obesity; Bulimia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided Self Help (Experimental): Guided Self Help intervention to reduce binge eating
  Interventions: Behavioral: Guided Self Help
- Treatment As Usual (Placebo Comparator): No intervention for binge eating (treatment as usual in the form of bariatric surgery)
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Guided Self Help — A behaviourally orientated guided self help book designed to reduce binge eating prior to surgery
  Arms: Guided Self Help
Other: Treatment As Usual — Binge eating disordered participants receive treatment as usual in the form of bariatric surgery (i.e. no pre-operative intervention to reduce binge eating)
  Arms: Treatment As Usual

SUMMARY:
To demonstrate the effectiveness of an easily administered intervention (guided self help) aimed at reducing binge eating in patients undergoing bariatric surgery.

The investigators hypothesize that patients who have guided self help pre-operatively will have reduced episodes of bingeing pre-operatively compared to those having treatment as usual (bariatric surgery), which will be maintained in the post-operative period, and will be associated with improved weight loss and psychological outcomes after surgery.

DETAILED DESCRIPTION:
Binge eating disorder (BED) is distressing and common in patients who present for treatment for obesity. Despite this, it is often undiagnosed. Patients who have bariatric surgery have improvements in their eating patterns, including binge eating. However there is variability in the degree of weight loss and post-operative complications following bariatric surgery, associated with disordered eating.

Guided self help for BED (GSH) is a treatment which, like bariatric surgery, is effective in reducing the number of binge episodes in people who binge eat. It is not known whether GSH prior to surgery, in patients undergoing bariatric surgery has any additional benefit for reducing bingeing, or improving weight loss in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI >28 kg/m2)
* Pursuing bariatric surgery

Exclusion Criteria:

* Any illnesses which make the patient unsuitable
* If the patient is taking any medication which makes them unsuitable
* If the patient is pregnant or breast feeding
* If the patient has donated blood in the last three months
* If the patient has a history of alcoholism or substance dependency within the last 5 years
* If the patient has a history of major haematological, renal, gastrointestinal, hepatic, respiratory, cardiovascular or psychiatric disease or other illness or use of any medications, including over the counter products, which, in the opinion of the investigators would either interfere with the study or potentially cause harm to the volunteer
* If the patient has any medical or psychological condition or social circumstances which would interfere with their ability to participate reliably in the trial
* If the patient is without access to a telephone
* If the patient is currently receiving or intends to receive treatment with an investigational drug within the next 2 months If the patient is currently receiving or intends to receive treatment for binge eating
* If the patient currently suffers with severe depression, as indicated by a Beck Depression Inventory Score greater than 28

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in body mass index point | baseline, pre-operatively, 3 month, 6 month and 1 year follow up

SECONDARY OUTCOMES:
Binge episodes | baseline, pre-operatively, 3 month, 6 month and 1 year follow up
  -Number of binge episodes per 28 days
Complication or reversal of surgery | 3 month, 6 month and 1 year follow up
  Surgical complication or reversal of bariatric surgery as per case notes
Quality of life | baseline, pre-operative, 3 month, 6 month and 1 year follow up
  Score on SF-36, IQoL-lite, Hospital anxiety and depression scale (HADS), and PANAS (positive and negative affect scale)
Eating behaviour | baseline, pre-operatively, 3 month, 6 month and 1 year follow up
  Emotional, externally driven, disinhibited, restrained eating patterns and weight and shape concerns as measured by Eating disorders examination questionnaire (EDE-Q), Dutch Eating Behaviour Questionnaire (DEBQ), Three factor eating questionnaire (TFEQ)
Drug and alcohol misuse | pre-operatively, baseline, 3 month, 6 month and 1 year follow up
  As measured by AUDIT drug and alcohol assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Scholtz, MRCPsych, Principal Investigator — Imperial College London
Locations (1):
- Obesity, Endocrine and Medical Clinics at Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The IPD has been shared with Prof. Alex Blakemore as planned, who was conducting the genetic part of the study and who is using the data in wider analysis.